CLINICAL TRIAL: NCT05452954
Title: A Non-randomized Pilot Study on Brief Behavioral Parent Training for Behavioral Problems of Children With ADHD Symptoms.
Brief Title: Psychosocial ADHD Interventions - Brief Parent Training
Acronym: PAINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Accare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METc 2020/459
Record Dates: First submitted 2022-06-01; First posted 2022-07-12 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: ADHD; ADHD - Combined Type; ADHD Predominantly Inattentive Type; ADHD, Predominantly Hyperactive-Impulsive Type; Behavior Problem; Behavioral Problem; Problem Behavior; Behavioral Symptoms; Child Behavior Problem; Disruptive Behavior
Keywords: behavioral parent training; brief behavioral parent training; first-line behavioral parent training; psychosocial ADHD intervention; parent training; first-line treatment ADHD; children 4-11 years
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Mental Disorders; Problem Behavior; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief behavioral parent training (Other): A newly developed, easily applicable, individually tailored first-line behavioral training for parents of children (4-12 years) with behavioral problems and (symptoms of) ADHD, that will be provided in an early stage, before other treatments have been applied.
  Interventions: Behavioral: Brief behavioral parent training

INTERVENTIONS:
Behavioral: Brief behavioral parent training — In the newly developed intervention, both stimulus control and contingency management techniques will be offered in a brief behavioral parent training consisting of two intervention sessions and one booster session.
  Other Names: paint-p; Psychosocial ADHD Interventions - Parent-training

SUMMARY:
This pilot study investigates a new, easily applicable, individually tailored first-line behavioral training for parents of children (4-12 years) with (symptoms of) ADHD, that will be provided in an early stage, before other treatments have been applied. In this pilot study the feasibility of the newly developed intervention will be evaluated by exploring program acceptability, including client satisfaction, recruitment, retention, treatment fidelity and therapist satisfaction. Also acceptability of potential outcome measures will be explored, including preliminary tests of efficacy.

DETAILED DESCRIPTION:
The study will be a non-randomized pilot study. The newly developed brief behavioral parent training has not been studied yet. Therefore, the current project aims at evaluating its feasibility. Furthermore, this project aims to explore whether parents' and their children's functioning improves from pre to post intervention. This will be assessed by investigating changes over time in the treatment group, and, if possible, by comparing these with changes in a control group that was included in a previous microtrial with an almost identical design and intervention.

OBJECTIVES

The primary objective of this study is evaluating the feasibility of the newly developed behavioral parent training This will be done by exploring its acceptability, including client satisfaction, recruitment, retention, treatment fidelity and therapist satisfaction. Furthermore, the acceptability of both primary and secondary outcome measures will be evaluated on a number of variables, such as frequency and duration of the assessment according to participants and response and completion rates. Preliminary tests of efficacy will be conducted by investigating changes over time in the treatment group, and, if possible, comparing all outcome measures with control data from a previous study that has an almost identical design.

METHODS

Design

Baseline measurement (all outcome measures) will be done one week before session 1 (T0). The primary outcome will be assessed one and three weeks after session 2 (T1 and T2). At T2, all other outcome measures will be assessed as well. Follow-up measurement (all outcome measures) will be done three weeks after the booster session (T3). Sessions and measurements are planned the same way as could be done in a future RCT.

Participants

Participants are parents of children between four up to and including eleven years old with behavioral problems and diagnosed with ADHD or at least four symptoms of ADHD according to DSM-5.

Treatment

The intervention consists of three sessions; two two-hours training sessions and a one-hour booster session. Treatment will take place in an outpatient child and adolescent mental health setting. Therapists will be well-trained in behavioral techniques and experienced in behavioral parent training for children with behavioral problems.

Outcome variables

To assess feasibility, the following outcome measures are investigated:

* Parent satisfaction (25 items)
* Parent-rated acceptability of primary and secondary outcome measures (7 descriptive items)
* Therapist satisfaction (short self-developed evaluation questionnaire)
* Treatment fidelity (audio records of sessions; percentage addressed session items)
* Recruitment (average number of included patients each month, number of patients meeting the inclusion criteria but not willing to participate)
* Retention rate (percentage study drop-out and percentage treatment drop-out)
* Response and completion rates on outcome measures (percentage of parents that responded at all timepoints, percentage of completed measures at all time-points)

For a preliminary test of efficacy, primary outcomes are daily ratings of four individually selected target behaviors. Secondary outcomes are:

* Inattentive, hyperactive and impulsive behaviors of the child (SWAN)
* Children's symptoms of oppositional defiant disorder (DBDRS)
* Disruptive problem behaviors of the child (ECBI)
* Impairment of the child (IRS)
* Parenting sense of competence (PSOC) See 'Outcomes Measures' for more details on all measures.

Statistics

For a preliminary test of efficacy, two research questions are formulated. The primary research question concerns the change from pre to post intervention within the treatment group. To analyze whether participants improve on daily ratings of problem behavior (primary outcome measure), a weekly mean-level will be derived on the basis of the daily ratings of the selected target behaviors in specific situations over five schooldays.

The secondary research question for preliminary efficacy concerns the comparison of the treatment group with historic controls. The change on primary and secondary outcome measures in the intervention group will be compared to the change in the historic control group.

Both research questions will be answered by a multilevel analysis (mixed modeling), which takes missing data into account. Three hierarchical levels will be distinguished: outcomes (level 1) nested within subjects (level 2), nested in therapists (level 3). A random intercept at therapist level will be included only if the Likelihood Ratio Test shows a significant improvement of the model fit. Condition (parent training vs control) will be inserted as between subjects factor and time (T1, T2, T3) as within subjects variable. To control for baseline differences, T0 scores will be inserted as fixed factor. As an historic control group will be used, also age, sex, ADHD symptoms (as measured by the SWAN) and ODD symptoms (as measured by the DBDRS) at T0 will be included, but only when groups differ on these variables at T0.

Data will be analyzed on an intention to treat basis. In all statistical analyses an alpha of 0.05 will be used.

Power analysis

A power analysis was executed for the primary pre-post within group analysis. Taking into account the lowest within condition effect size found in a previous study on brief behavioral parent training (d=.57), an effect size of f=.285 (f=d/2) is assumed for this power analysis. Given alpha=.05 and power 1-β=.80, a total number of 28 study participants will be required.

ELIGIBILITY:
Inclusion Criteria:

* A) The child is diagnosed with ADHD according to DSM-5 as measured by the Parent Interview for Child Symptoms [PICS] and the Teacher Telephone Interview [TTI] or; B) The child has at least four impairing symptoms of ADHD (at least four symptoms of ADHD as measured by the Parent Interview for Child Symptoms [PICS] and at least two symptoms measured by the Teacher Telephone Interview [TTI]; and significant impairment rated >3 on the Impairment Rating Scale [IRS]).
* The child is between four up to and including eleven years old and is attending a Dutch primary school.
* The child has an IQ higher than 70. If an IQ-score is not available, this will be estimated with two subtests of the Wechsler Intelligence Scale for Children-V (Dutch edition; WISC-V-NL) or the Wechsler Preschool and Primary Scale of Intelligence-III (Dutch edition; WPSSI-III-NL).
* Parents/caregivers have given their informed consent for participation.

Exclusion Criteria:

* Parents received behavioral parent training (individual or group) aimed at ADHD or behavioral problems of the child in the past year.
* The child is currently taking psychotropic medication or has taken psychotropic medication in the past month.
* The child has a DSM-5 or a DSM-IV-TR based diagnosis of an Autism Spectrum Disorder.
* There are problems with the child and/or the family that require immediate intensive intervention (e.g., crisis in the family).
* The child does not live in one household during weekdays.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Change in daily ratings of target behaviors by ecological momentary assessment | T0 (baseline) 1 week before intervention; T1 (post-training 1) 1 week after intervention session 2; T2 (post-training 2) 3 weeks after intervention session 2; T3 (follow-up) 3 weeks after intervention booster session.
  The primary outcome measure will be daily ratings of 4 selected target behaviors. The target behaviors will be selected from a list of 31 problem behaviors on which parents indicate whether these behaviors daily occur (yes/no). For the items scored as yes parents rate the severity of the behaviors on a 5-point Likertscale ranging from 1 not severe to 5 extremely severe. Parents will be asked to choose 4 target behaviors from this list (i.e. the behaviors that they prefer to work on in the training). They will also be asked to specify in which situations these behaviors typically occur. During a week (5 schooldays), a member of the research team will make daily phone calls with participating parents to evaluate whether the 4 selected target behaviors occurred in the past 24 hours (yes/no). Items scored as No will be rated 0, items scored as Yes will be rated on a 5-point Likertscale ranging from 1 not severe to 5 extremely severe (daily score min = 0, max = 20).

SECONDARY OUTCOMES:
Change in inattentive, hyperactive and impulsive behaviors of the child. | T0 (baseline) 1 week before intervention; T2 (post-training) 3 weeks after intervention session 2; T3 (follow-up) 3 weeks after intervention booster session
  Symptoms of inattentiveness, hyperactivity and impulsivity will be assessed by the Strengths and Weaknesses of ADHD symptoms and Normal behavior rating scale (SWAN). The SWAN is a list containing 18 items measuring inattentive, hyperactive, and impulsive behaviors. The SWAN is based on an earlier scale, the Swanson, Nolan and Pelham Teacher and Parent (SNAP) Rating Scale. It consists of 18 items, rated on a 7-point scale ranging from -3 'far below average' to 3 'far above average' (min = -54, max = 54). Reliability and validity have both been evaluated as adequate.
Change in children's symptoms of oppositional defiant disorder | T0 (baseline) 1 week before intervention; T2 (post-training) 3 weeks after intervention session 2; T3 (follow-up) 3 weeks after intervention booster session
  A subscale (8 items) of the Dutch version of the Disruptive Behavior Disorder Rating Scales (DBDRS) will be used to identify symptoms of oppositional defiant disorder (ODD). The DBDRS has been designed to assess symptoms of externalizing disorders that can be completed by parents or teachers. The parent/caregiver is asked to indicate the degree to which a statement describes their child's behavior. Responses include; 'not at all' (0), 'just a little' (1), 'pretty much' (2), and 'very much' (3) (min = 0, max = 24). The subscale ODD has good construct validity and internal consistency (α = .88).
Change in disruptive problem behaviors of the child | T0 (baseline) 1 week before intervention; T2 (post-training) 3 weeks after intervention session 2; T3 (follow-up) 3 weeks after intervention booster session
  Children's current disruptive problem behaviors will be assessed by the Dutch version of the Eyberg Child Behavior Inventory (ECBI). The ECBI is a 36-item questionnaire for parents of children aged 2 to 16, consisting of two scales. The intensity scale measures the frequency of specific problem behavior on a 7-point Likert scale (1=never to 7=always, min = 36, max = 252). On the problem scale, parents report whether the specific behavior-item is problematic for parents or not on a dichotomous scale (0=no, 1=yes; min = 0, max = 36). Psychometric qualities (internal consistency, test-retest reliability and validity) of the Dutch version of the ECBI are good.
Change in impairment of the child | T0 (baseline) 1 week before intervention; T2 (post-training) 3 weeks after intervention session 2; T3 (follow-up) 3 weeks after intervention booster session
  Impairment of the child will be assessed with the Impairment Rating Scale (IRS). The IRS measures impairment on seven domains, including relationships with peers, siblings, and parents, family functioning, academic progress, self-esteem, and overall impairment. Caregivers are asked to score how impaired they think their child is in each domain, from 0 'no problem' to 6 'extreme problem' (min = 0, max = 42). The IRS has been demonstrated to validly identify impairment in children with ADHD, with a score of 3 or more indicating clinically significant impairment.
Change in parenting sense of competence | T0 (baseline) 1 week before intervention; T2 (post-training) 3 weeks after intervention session 2; T3 (follow-up) 3 weeks after intervention booster session
  The subscale Efficacy of the Parenting Sense of Competence Scale (PSOC) will be used to measure parenting self-efficacy. It contains 8 items (e.g., 'Being a parent is manageable, and any problems are easily solved') on which parents have to indicate their level of agreement. Ratings have to be made on a 6-point scale, ranging from 1 'strongly agree' to 6 'strongly disagree' (min = 8, max = 42). Good internal consistency and construct validity have been reported.

OTHER OUTCOMES:
Parent satisfaction | T3 (follow-up) 3 weeks after intervention booster session
  Parent satisfaction and acceptability of the intervention will be measured using an evaluation questionnaire containing 25 items about parental satisfaction and usefulness of training parts, the ease with which parents can combine the training with daily life, the use of learned skills, the perceived influence on their child's behavior, perceived helpfulness of the training, and whether parents would recommend the training to other parents.
  The parent satisfaction questionnaire used in this study is based on the Parent Satisfaction Questionnaire and the Therapy Attitude Inventory. Ratings are made on a 5-point scale, ranging from 1 'totally disagree' to 5 'totally agree' (min = 25, max = 125).
Parent-rated acceptability of outcome measures | T3 (follow-up) 3 weeks after intervention booster session
  Acceptability of primary and secondary measures according to participants will be measured using seven self-developed evaluation questions on frequency and duration of measurements, analyzed on item level. Ratings are made on a 5-point scale, on each item ranging from min=1 (too few/ too short/ strongly disagree) to max=5 (too much/ too long/ strongly agree).
Therapist satisfaction | Through study completion, an average of 1,5 year.
  Therapists' satisfaction will be measured after inclusion has finished, using a short self-developed evaluation questionnaire on acceptability and usefulness of the intervention according to therapists, analyzed on item level. Ratings are made on a 5-point scale, on each item ranging from min=1 (too few/ too short/ strongly disagree) to max=5 (too much/ too long/ strongly agree).
Treatment fidelity | Through study completion, an average of 1,5 year.
  Therapists will be asked to make audio records of each session and score a treatment fidelity checklist after each session. The percentage of addressed session items in each session will be checked in two ways; through the session-forms from the therapists, and through scoring the selected audiotapes (20% of the sessions, randomly selected).
Retention rate | Through study completion, an average of 1,5 year.
  The number of parents dropped out from the study and from the treatment will be reported.
Response and completion rate | Through study completion, an average of 1,5 year.
  The percentage of parents that responded at all timepoints will be reported, as welll as the percentage of completed measures at all timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: B. J. Van den Hoofdakker, Prof. dr., Principal Investigator — Accare
Locations (1):
- Accare, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Hoofdakker BJ, van der Veen-Mulders L, Sytema S, Emmelkamp PMG, Minderaa RB, Nauta MH. Effectiveness of behavioral parent training for children with ADHD in routine clinical practice: a randomized controlled study. J Am Acad Child Adolesc Psychiatry. 2007 Oct;46(10):1263-1271. doi: 10.1097/chi.0b013e3181354bc2. PMID 17885567
- [Background] Swanson JM, Schuck S, Porter MM, Carlson C, Hartman CA, Sergeant JA, Clevenger W, Wasdell M, McCleary R, Lakes K, Wigal T. Categorical and Dimensional Definitions and Evaluations of Symptoms of ADHD: History of the SNAP and the SWAN Rating Scales. Int J Educ Psychol Assess. 2012 Apr;10(1):51-70. PMID 26504617
- [Background] Swanson, J. M. (1992). School-based assessments and interventions for ADD students. Irvine, CA: KC Publishing.
- [Background] Lakes KD, Swanson JM, Riggs M. The reliability and validity of the English and Spanish Strengths and Weaknesses of ADHD and Normal behavior rating scales in a preschool sample: continuum measures of hyperactivity and inattention. J Atten Disord. 2012 Aug;16(6):510-6. doi: 10.1177/1087054711413550. Epub 2011 Aug 1. PMID 21807955
- [Background] Oosterlaan, J., Baeyens, D., Scheres, A., Antrop, I., Roeyers, H., & Sergeant, J. (2008). VvGK6-16: Vragenlijst voor gedragsproblemen bij kinderen 6 tot en met 16 jaar. Amsterdam: Pearson.
- [Background] Pelham WE Jr, Gnagy EM, Greenslade KE, Milich R. Teacher ratings of DSM-III-R symptoms for the disruptive behavior disorders. J Am Acad Child Adolesc Psychiatry. 1992 Mar;31(2):210-8. doi: 10.1097/00004583-199203000-00006. PMID 1564021
- [Background] Eyberg, S. M., & Pincus, D. (1999). ECBI & SESBI-R: Eyberg child behavior inventory and sutter-eyberg student behavior inventory-revised: Professional manual. Lutz, Florida: Psychological Assessment Resources.
- [Background] van der Veen-Mulders L, Hoekstra PJ, Nauta MH, van den Hoofdakker BJ. Preschool children's response to behavioural parent training and parental predictors of outcome in routine clinical care. Clin Psychol Psychother. 2018 Jan;25(1):1-9. doi: 10.1002/cpp.2117. Epub 2017 Aug 30. PMID 28857440
- [Background] Weeland J, van Aar J, Overbeek G. Dutch Norms for the Eyberg Child Behavior Inventory: Comparisons with other Western Countries. J Psychopathol Behav Assess. 2018;40(2):224-234. doi: 10.1007/s10862-017-9639-1. Epub 2017 Dec 2. PMID 29937620
- [Background] Abrahamse ME, Junger M, Leijten PH, Lindeboom R, Boer F, Lindauer RJ. Psychometric Properties of the Dutch Eyberg Child Behavior Inventory (ECBI) in a Community Sample and a Multi-Ethnic Clinical Sample. J Psychopathol Behav Assess. 2015;37(4):679-691. doi: 10.1007/s10862-015-9482-1. Epub 2015 Mar 25. PMID 26640320
- [Background] Fabiano GA, Pelham WE Jr, Waschbusch DA, Gnagy EM, Lahey BB, Chronis AM, Onyango AN, Kipp H, Lopez-Williams A, Burrows-Maclean L. A practical measure of impairment: psychometric properties of the impairment rating scale in samples of children with attention deficit hyperactivity disorder and two school-based samples. J Clin Child Adolesc Psychol. 2006 Sep;35(3):369-85. doi: 10.1207/s15374424jccp3503_3. PMID 16836475
- [Background] Gibaud-Wallston, J., & Wandersman, L. P. (1978). Development and utility of the parenting sense of competence scale. Paper presented at the Annual Meeting of the American Psychological Association, Toronto.
- [Background] Johnston, C., & Mash, E. J. (1989). A measure of parenting satisfaction and efficacy. Journal of Clinical Child Psychology, 18(2), 167-175. doi:10.1207/s15374424jccp1802_8
- [Background] van der Veen-Mulders L, Hoekstra PJ, Nauta MH, van den Hoofdakker BJ. Are parental changes related to improvements in preschool children's disruptive behaviours? Clin Psychol Psychother. 2020 Jan;27(1):24-33. doi: 10.1002/cpp.2402. Epub 2019 Dec 4. PMID 31614051
- [Background] Gilmore L, Cuskelly M. Factor structure of the Parenting Sense of Competence scale using a normative sample. Child Care Health Dev. 2009 Jan;35(1):48-55. doi: 10.1111/j.1365-2214.2008.00867.x. Epub 2008 Oct 22. PMID 18991983
- [Background] Ohan, J. L., Leung, D. W., & Johnston, C. (2000). The parenting sense of competence scale: Evidence of a stable factor structure and validity. Canadian Journal of Behavioural Science / Revue Canadienne Des Sciences Du Comportement, 32(4), 251-261. doi:10.1037/h0087122
- [Background] Bearss K, Johnson C, Handen B, Smith T, Scahill L. A pilot study of parent training in young children with autism spectrum disorders and disruptive behavior. J Autism Dev Disord. 2013 Apr;43(4):829-40. doi: 10.1007/s10803-012-1624-7. PMID 22941342
- [Background] Eyberg, S. M. (1993). Consumer satisfaction measures for assessing parent training programs. In L. VandeCreek, S. Knapp & T. L. Jackson (Eds.), (pp. 377-382). Sarasota, FL: Professional Resource Press/Professional Resource Exchange. Retrieved from http://search.ebscohost.com.proxy-ub.rug.nl/login.aspx?direct=true&db=psyh&AN=1994-97027-025&site=ehost-live&scope=site
- [Background] Eyberg SM, Johnson SM. Multiple assessment of behavior modification with families: effects of contingency contracting and order of treated problems. J Consult Clin Psychol. 1974 Aug;42(4):594-606. doi: 10.1037/h0036723. No abstract available. PMID 4847264
- [Background] APA. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Arlington, VA: American Psychiatric Association.
- [Background] Hornstra R, van der Oord S, Staff AI, Hoekstra PJ, Oosterlaan J, van der Veen-Mulders L, Luman M, van den Hoofdakker BJ. Which Techniques Work in Behavioral Parent Training for Children with ADHD? A Randomized Controlled Microtrial. J Clin Child Adolesc Psychol. 2021 Nov-Dec;50(6):888-903. doi: 10.1080/15374416.2021.1955368. Epub 2021 Aug 23. PMID 34424102
- [Background] Twisk J, de Boer M, de Vente W, Heymans M. Multiple imputation of missing values was not necessary before performing a longitudinal mixed-model analysis. J Clin Epidemiol. 2013 Sep;66(9):1022-8. doi: 10.1016/j.jclinepi.2013.03.017. Epub 2013 Jun 21. PMID 23790725